CLINICAL TRIAL: NCT05753306
Title: A Phase II Study of Robotic Cytoreduction and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Patients With Gastric Cancer and Limited Peritoneal Metastasis: ROBO-CHIP Trial
Brief Title: Robotic Cytoreduction and Hyperthermic Intraperitoneal Chemotherapy for Treatment of Gastric Cancer With Limited Peritoneal Metastasis, ROBO-CHIP Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-004680; NCI-2023-00431 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-004680 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Metastatic Malignant Neoplasm in the Peritoneum
MeSH Terms: interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gastrectomy; Magnetic Resonance Spectroscopy; Paclitaxel; taxane; Taxes; Albumin-Bound Paclitaxel; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (gastrectomy, HIPEC) (Experimental): Patients undergo collection of stool and blood sample before and after surgery. Patients also undergo robotic gastrectomy and HIPEC with docetaxel and cisplatin on study. Patients undergo CT, MRI, or PET/CT scans throughout the trial.
  Interventions: Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Gastrectomy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Drug: Paclitaxel; Drug: Hyperthermic Intraperitoneal Chemotherapy

INTERVENTIONS:
Drug: Cisplatin — Given via HIPEC
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Gastrectomy — Undergo robotic gastrectomy
  Other Names: Gastric Resection
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PE/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Complete questionnaire
Drug: Paclitaxel — Given via HIPEC
  Other Names: Taxane; Taxol; 5beta,20-Epoxy-1,2-alpha,4,7beta,10beta,13alpha-hexahydroxytax-11-en-9-one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)-N-benzoyl-3-phenylisoserine; Taxol Konzentrat; Praxel; Abraxane; Naveruclif; Pazenir
Drug: Hyperthermic Intraperitoneal Chemotherapy — Undergo HIPEC
  Other Names: HIPEC

SUMMARY:
This phase II clinical trial tests how well robotic cytoreduction and hyperthermic intraperitoneal chemotherapy (HIPEC) in treating patients with gastric cancer that has spread to the tissue that lines the wall of the abdominal cavity (peritoneum). Gastric cancer is the third leading cause of cancer related deaths worldwide and peritoneal metastasis are found in 30% of patients at time of diagnosis. Patients with peritoneal metastasis have poor survival rates. Traditional surgery is done with a large incision and has a high complication rate and longer hospital stays. Robot assisted (robotic) cytoreduction is a surgical option that uses small incisions and there is less risk of complications. HIPEC involves infusing heated chemotherapy into the abdominal cavity during surgery. Robotic cytoreduction together with HIPEC may improve recovery and decrease complications after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Restricted to 18 to 80 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Histologic confirmation of gastric adenocarcinoma including all subtypes and Siewert type II/III gastroesophageal (GE) junction adenocarcinomas
* Absolute neutrophil count >= 1,500 / uL
* Platelets >= 50,000 / Ul
* Serum creatinine <= 1.5 mg / dL
* Adequate nutritional status (Albumin >= 3.5)
* Metastasis confined to the peritoneum:

  * Positive peritoneal cytology
  * Peritoneal metastasis on diagnostic laparoscopy
  * Peritoneal metastasis on imaging
* Response to systemic chemotherapy defined as at least one of the following:

  * Reduction (>= 30%) in standardized uptake value (SUV) max [Response Evaluation Criteria in Solid Tumors (RECIST) criteria]
  * Reduction in size of primary tumor, regional lymph node or peritoneal metastasis on imaging (>= 20% decrease in the longest diameter of target lesion) RECIST criteria
  * Reduction ( >= 30%) in Peritoneal Carcinomatosis Index (PCI) or conversion of peritoneal cytology
  * Reduction ( >= 30%) in serum tumor markers CEA or CA 19-9
* Peritoneal Carcinomatosis Index (PCI) =< 7 and surgeon deems high likelihood for a complete cytoreduction
* Body Mass Index (BMI) =< 35 kg/m^2

Exclusion Criteria:

* Distant metastatic disease not limited to peritoneum, such as solid organ metastases (liver, lung, bone, distant lymph node, etc)
* Malignant ascites at time of study enrollment
* Comorbidities that would preclude protocol therapy
* Subjects deemed unable to comply with study and/or follow-up procedures
* Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | Up to 30 days post-surgery
  Recorded as number of days in hospital following surgery.
30 day readmission rate | Up to 30 days post-surgery
  Assessed by the number of participants who are re-admitted to the hospital after being discharged post-surgery
Adverse Events | Up to 30 days post surgery
  Assessed by Clavien-Dindo Classification (grade 1-5, grade 1 being least severe and grade 5 being death)

SECONDARY OUTCOMES:
Operative time | Intraoperative
  Recorded as the time from incision to close
Opioid consumption | Up to 42 months
  Assessed by morphine milligram equivalents during hospitalization and post-surgical recovery.
Nursing reported pain scores | Up to 42 months
  As recorded (mean and max) during hospitalization and post-surgery follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Travis E Grotz, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials